CLINICAL TRIAL: NCT06529666
Title: MRWeight: Medical Residents Learning Weight Management Counseling Skills -- A Multi-Modal, Technology-Assisted, Spaced Education Program
Brief Title: Medical Residents Learning Weight Management Counseling Skills
Acronym: MRWeight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Albert Einstein College of Medicine (Other); Penn State University (Other); The Methodist Hospital Research Institute (Other); Boston University (Other); Stanford University (Other); Temple University (Other); University of California, Davis (Other); Stony Brook University (Other)
Responsible Party: Principal Investigator, Rajani Sadasivam, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00000691; 1R01DK134372-01 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Weight Management Counseling
Keywords: weight management counseling; Internship and Residency; skills and adoption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison Arm (Active Comparator): Residents in comparison arm receive a core foundation course and will take part in all 3 assessments (including 3 surveys and 2 video communication assessments) over the course of 18 months.
  Interventions: Behavioral: PowerPoint of the foundational course
- Intervention Arm (Experimental): Residents in the intervention arm will receive (in addition to the core foundation course) 6 email modules and practice video communication assessments on weight management counseling. They will also attend 2 educational session and take part in all 3 assessments (including 3 surveys and 2 video communication assessments) over the course of 18 months.
  Interventions: Behavioral: Didatic Session 1: Core Foundation Course; Behavioral: The 3Ps Program; Behavioral: Didactic session 2; Behavioral: Email reinforcement; Behavioral: PowerPoint of the foundational course

INTERVENTIONS:
Behavioral: Didatic Session 1: Core Foundation Course — A 45-minute foundational presentation covering key Weight Management Counseling (WMC) concepts, obesity bias, and cultural humility facilitated by a trained clinician-educator at the residency program delivered at baseline.
  Arms: Intervention Arm
Behavioral: The 3Ps Program — 6 email modules delivered over months 2-8). Each 3P module will allow the resident to:
  (1) Prepare: Review relevant concepts and demonstration videos sent via an email to prepare for completing the VCA vignettes; (2) Practice: Respond to brief vignettes of various 5As WMC challenging scenarios by audio recording their spoken response on the VCA tool; and (3) Process: Reflect on actionable expert and crowdsourced analogue patient feedback on the quality of their responses to each VCA vignette.
  Arms: Intervention Arm
Behavioral: Didactic session 2 — (months 8-10): This 45-minute session will discuss key barriers to WMC adoption in clinical practice using real-world cases captured from residents facilitated by a trained clinician-educator at the residency program.
  Arms: Intervention Arm
Behavioral: Email reinforcement — 2 emails in months 10-12 covering key concepts in the preceding components.
  Arms: Intervention Arm
Behavioral: PowerPoint of the foundational course — Residents will receive a core foundation slides on weight management counselling

SUMMARY:
The goal of this study is to addresses the lack of weight management training physicians receive during their residency training. The main questions it aims to answer are:

* How affective is the MRWeight curriculum at increasing medical residents weight management counseling (WMC) skills.
* Evaluate residents' adoption of WMC skills in encounters with their patients
* what would be the best way to get residents to adopt the WMC skills Residents in the comparison group will receive a course on obesity and weight management. The residents in the intervention group will have to attend 2 informational sessions and will receive 6 email modules on WMC. Both groups will also take part in 3 assessments over the course of 18 months to see which group has better WMC skills.

DETAILED DESCRIPTION:
Overweight and obesity have reached epidemic proportions in the United States, proving to be a very difficult health challenge for both patients and the physicians who care for them. Excess weight is a major contributor to heart disease, stroke, and type 2 diabetes. Addressing overweight and obesity in clinical visits is critical to treating and preventing these obesity-associated diseases. However, Weight Management Counseling (WMC) uptake is low, and physicians report lack of training as a critical barrier to WMC. Residency training is a crucial time to influence physicians' current and future practice, yet there is no evidence-supported WMC curriculum for residents. Informed by two pilot studies, MRWeight will use spaced-education to train residents to deliver WMC using the 5As framework (Ask, Advise, Assess, Assist, Arrange) and patient-centered counseling. As such, MRWeight will be delivered in short segments and spaced over 12 months using four components: didactic session 1 - a discussion of WMC foundational concepts; 3Ps program (Prepare, Practice, Process) - an email program using the Video-based Communication Assessment (VCA) to facilitate practice of challenging cases; didactic session 2 - a discussion of key barriers to practicing WMC; and email reinforcement of concepts covered in the preceding components. Each component, guided by Social Cognitive Theory (SCT), is designed to build on and reinforce the training provided by the other components. Using a pair-matched group randomized controlled trial (RCT) including 8 Internal Medicine residency programs, we will test the MRWeight intervention with 3 cohorts of postgraduate year 1 residents followed for 18 months. Comparison arm residents will be emailed the PowerPoint of a foundational course on WMC, but unlike those in the Intervention, comparison sites will not include the didactic sessions or the 3Ps program. Our aims are: Aim 1 will evaluate the effectiveness of the MRWeight Intervention for increasing residents' WMC skills at 12 months; Aim 2 will evaluate residents' self-reported adoption of WMC skills in their encounters with patients in clinical practice at 18 months; Aim 3 will explore possible mechanisms (mediators) and moderators of the intervention's effect on Aim 1 and 2 outcomes (residents' WMC skills and adoption). The study will be the first large trial to test a curriculum that has been integrated into Internal Medicine residency programs for teaching WMC skills. The multi-PIs (Drs. Ockene and Sadasivam) will build on 36-years of successfully conducting large randomized trials to evaluate training programs, including those that taught the 5As and patient-centered counseling for WMC, in 18 medical schools, 10 residency sites, and 10 primary care settings. This study is timely, given public health momentum strongly advocating for physician training and involvement in WMC and the dissemination and implementation of clinical guidelines for obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

* All PGY1 residents in participating sites

Inclusion Criteria for participating site:

* The program is willing and able to incorporate the MRWeight program into the PGY1 core curriculum.
* The residency director will allow PGY1s to complete surveys and curriculum evaluations online or in class and to complete a standardized assessment of their knowledge and use of WMC, and
* The site will allow inclusion of three successive cohorts of PGY1s to ensure more than a sufficient number of residents to adequately test the effect of the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
WMC skills VCA (video Communications assessment) assessment | Completed during month 1 and again at month 12 post recruitment.
  Residents in both arms will be asked to complete the assessment VCA vignettes that will include a series of vignettes representing challenging cases. 4-6 trained raters blinded to the residents' study arm (intervention vs. comparison) will rate the residents' responses.
Change in WMC skills assessment | Completed during months 1, 12 and 18 post recruitment.
  This measure will be assessed using an online survey at baseline (study start), at 12 months, and 18 months.

SECONDARY OUTCOMES:
Change in adoption scale Scores at eighteen months | Completed during months 1, 12 and 18 post recruitment.
  This measure will be assessed using Adoption scale (7-item checklist assessing resident adoption of WMC skills in their encounters with patients in clinical practice) on a 5-point on a Likert Scale [never (0) to always (4)].

CONTACTS AND LOCATIONS:
Overall Officials: RAJANI SADASIVAM, PhD, Principal Investigator — UMass Chan Medical School
Locations (8):
- United States (8):
  - Stanford University, Palo Alto, California
  - UC Davis, Sacramento, California
  - Boston University, Boston, Massachusetts
  - Stony Brook, East Setauket, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Penn State University, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No